CLINICAL TRIAL: NCT06771154
Title: Adebrelimab Plus Carboplatin/Paclitaxel Followed by Adebelizumab with or Without Apatinib in the Treatment of Advanced Recurrent/Metastatic Endometrial Cancer (A-CAPE): a Multicenter, Randomized, Controlled, Open-Label Clinical Trial
Acronym: A-CAPE
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PekingUMCH-EC(A-CAPE)
Record Dates: First submitted 2025-01-08; First posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2024-12

CONDITIONS: Recurrent/Metastatic Endometrial Cancer
Keywords: Recurrent/Metastatic Endometrial Cancer; Adebrelimab; Apatinib; PD-L1; maintenance immune-targeted combination therapy
MeSH Terms: conditions — Endometrial Neoplasms | interventions — apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Maintenance Therapy Group with Adebrelimab Combined with Apatinib (Experimental): Chemotherapy Phase (Total of 6 cycles, each cycle 21 days) Carboplatin AUC 5 mg/mL/min, administered on the first day of each cycle; Paclitaxel 175 mg/m², intravenous infusion for 3 hours, administered on the first day of each cycle; Adebelimab: Fixed dose of 1200 mg per administration, on the first day of each cycle, until the end of chemotherapy or until treatment is discontinued due to disease progression, intolerable toxicity, or other reasons specified in the protocol.
  Maintenance Therapy Phase (Each cycle 21 days) Adebelizumab: Fixed dose of 1200 mg per administration, IV (intravenous), Q3W (every 3 weeks), on the first day of each cycle, for a maximum of two years; Apatinib: 250 mg, once daily (qd), orally (po); Treatment continues until disease progression, intolerable toxicity, or other reasons specified in the protocol result in discontinuation.
  Interventions: Drug: Adebelimab Combined with Apatinib
- Maintenance Therapy Group with Adebrelimab (Active Comparator): Chemotherapy Phase (Total of 6 cycles, each cycle 21 days) Carboplatin AUC 5 mg/mL/min, administered on the first day of each cycle. Paclitaxel 175 mg/m², intravenous infusion for 3 hours, administered on the first day of each cycle. Adebelimab, Fixed dose of 1200 mg per administration, on the first day of each cycle, until the end of chemotherapy or until treatment is discontinued due to disease progression, intolerable toxicity, or other reasons specified in the protocol.
  Maintenance Therapy Phase (Each cycle 21 days) Adebelizumab, Fixed dose of 1200 mg per administration, IV (intravenous), Q3W (every 3 weeks), on the first day of each cycle, for a maximum of two years.
  Treatment continues until disease progression, intolerable toxicity, or other reasons specified in the protocol result in discontinuation.
  Interventions: Drug: Adebelimab

INTERVENTIONS:
Drug: Adebelimab Combined with Apatinib — Chemotherapy Phase (Total of 6 cycles, each cycle 21 days) Carboplatin AUC 5 mg/mL/min, administered on the first day of each cycle. Paclitaxel 175 mg/m², intravenous infusion for 3 hours, administered on the first day of each cycle.
  Adebelizumab, Fixed dose of 1200 mg per administration, on the first day of each cycle, until the end of chemotherapy or until treatment is discontinued due to disease progression, intolerable toxicity, or other reasons specified in the protocol.
  Maintenance Therapy Phase (Each cycle 21 days) Adebelimab, Fixed dose of 1200 mg per administration, IV (intravenous), Q3W (every 3 weeks), on the first day of each cycle, for a maximum of two years; Apatinib, 250 mg, once daily (qd), orally (po). Treatment continues until disease progression, intolerable toxicity, or other reasons specified in the protocol result in discontinuation.
  Arms: Maintenance Therapy Group with Adebrelimab Combined with Apatinib
Drug: Adebelimab — Chemotherapy Phase (Total of 6 cycles, each cycle 21 days) Carboplatin AUC 5 mg/mL/min, administered on the first day of each cycle. Paclitaxel 175 mg/m², intravenous infusion for 3 hours, administered on the first day of each cycle.
  Adebelizumab, Fixed dose of 1200 mg per administration, on the first day of each cycle, until the end of chemotherapy or until treatment is discontinued due to disease progression, intolerable toxicity, or other reasons specified in the protocol.
  Maintenance Therapy Phase (Each cycle 21 days) Adebelimab, Fixed dose of 1200 mg per administration, IV (intravenous), Q3W (every 3 weeks), on the first day of each cycle, for a maximum of two years; Treatment continues until disease progression, intolerable toxicity, or other reasons specified in the protocol result in discontinuation.
  Arms: Maintenance Therapy Group with Adebrelimab

SUMMARY:
This study takes investigator-assessed Progression-Free Survival (PFS) as the primary endpoint, with plans to enroll 140 patients with advanced recurrent/metastatic endometrial cancer in a 1:1 ratio, randomized into an experimental group and a control group. The aim is to evaluate the efficacy and safety of Adebelimab (PD-L1) combined with Carboplatin/Paclitaxel treatment, followed by maintenance therapy with or without Apatinib in patients with advanced recurrent/metastatic endometrial cancer. Additionally, based on molecular testing results, the study will explore the PFS and Overall Survival (OS) of patients with Deficient Mismatch Repair/Microsatellite Instability-High(dMMR/MSI-H) and Proficient Mismatch Repai/Microsatellite Stability (pMMR/MSS) endometrial cancer, providing new precision treatment options for patients with recurrent and metastatic endometrial cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Histologically or cytologically confirmed diagnosis of primary advanced (FIGO stage III/IV) endometrial cancer patients, or first recurrent endometrial cancer with low likelihood of cure through radiotherapy, surgery, or a combination of both.
* Pathological type is not limited (excluding sarcomas for all pathological types).
* MMR/MSI test report available, or tumor tissue for MMR/MSI status testing can be provided.
* Patients with endometrial cancer who have not received systemic antitumor therapy or have ≤1 line of recurrence (including neoadjuvant, postoperative adjuvant chemotherapy, and concurrent chemotherapy), or have relapsed after completing systemic antitumor therapy with PD ≥ 6 months (limited to first recurrence).
* Discontinuation interval of ≥4 weeks for previous radiotherapy, chemotherapy, or hormone therapy; for patients who have failed platinum-based chemotherapy, a platinum-free interval of ≥6 months is required.
* ECOG score: 0-2, with an expected survival of ≥6 months.
* Patients have good organ function: without having received blood products, granulocyte colony-stimulating factor, interleukin-11, thrombopoietin, or thrombopoietin receptor agonists within 14 days prior to the first administration of the treatment drug in this protocol.Neutrophil count ≥ 1.5 × 10^9/L; Platelet count ≥ 80 × 10^9/L; Hemoglobin ≥ 80 g/L; Albumin ≥ 28 g/L; Total bilirubin ≤ 1.5 times the upper limit of normal (ULN); ALT, AST ≤ 3 times ULN (without liver metastasis) or ≤ 5 times ULN (in case of liver metastasis); Serum creatinine ≤ 1.5 times ULN; Coagulation function requirements: International Normalized Ratio (INR) ≤ 1.5 times ULN, Prothrombin Time (PT) ≤ 1.5 times ULN, Activated Partial Thromboplastin Time (APTT) ≤ 1.5 times ULN; Corrected serum electrolytes within normal range.
* Thyroid function: Thyroid-Stimulating Hormone (TSH) level ≤ 1 × ULN, or if TSH is not within the normal range, Free T4 ≤ 1 × ULN.
* Fertile women must undergo a pregnancy test (serum or urine) within 7 days prior to enrollment with a negative result and agree to use appropriate contraception during the trial period and for 3 months after the last dose of the investigational drug.
* Signed a written informed consent form and expected to have good compliance with the study protocol.

Exclusion Criteria:

* Individuals with known allergy or severe allergic reactions to the study drug or any of its excipients.
* Prior treatment with immune checkpoint inhibitors, including but not limited to other anti-PD-1 and anti-PD-L1 antibodies; prior treatment with small molecule anti-angiogenic targeted drugs (TKIs).
* Presence of other non-curable malignant tumors, except for those that have been definitively cured or locally curable cancers, such as skin basal or squamous cell carcinoma, cervical carcinoma in situ, or breast carcinoma in situ.
* Primary malignant tumors of the central nervous system, meningeal metastases, symptomatic brain metastases, or newly diagnosed and untreated brain metastases.
* Receipt of the following medications or treatments prior to the first dose of the study drug. Major surgery or trauma within 6 weeks with incomplete recovery (tissue biopsy for diagnostic purposes and procedures such as peripherally inserted central catheter [PICC] placement or port-a-cath implantation are allowed). Requirement for continuous high-dose systemic corticosteroids (>10 mg/day of prednisone or equivalent) or other systemic immunosuppressants (including but not limited to cyclophosphamide, azathioprine, methotrexate, thalidomide, tacrolimus, cyclosporine, mycophenolate mofetil, antithymocyte globulin, anti-tumor necrosis factor drugs), and the need for continued treatment after enrollment. [Note]: Topical, ocular, intra-articular, intranasal, and inhaled corticosteroids are allowed.
* History of severe infection within 90 days, such as severe pneumonia requiring hospitalization, bacteremia, infectious complications, etc.; active tuberculosis, patients with positive hepatitis B surface antigen (HBsAg+) and/or positive hepatitis B core antibody (HBcAb+) require hepatitis B virus deoxyribonucleic acid (HBV DNA) testing; if HBV DNA copy number is <1000 cps/mL or below the lower limit of detection at the research center, they may participate in the study and use anti-HBV drugs as prescribed, patients with positive hepatitis C virus antibody (HCV Ab+) require HCV RNA testing. HCV RNA-negative (defined as below the lower limit of detection at the research center) may participate in the study; human immunodeficiency virus (HIV) infection (anti-HIV positive).
* Receipt of first-line or second-line anti-cancer drug treatment within 4 weeks prior to the first dose; receipt of systemic treatment with herbs or immunomodulatory drugs (including thymosin, interferon, interleukin, excluding local use for pleural effusion control) with anti-cancer indications within 2 weeks prior to the first dose.
* Clinically significant cardiovascular disease, including but not limited to:

Diagnosis of deep venous thrombosis or pulmonary embolism within 1 month prior to the first dose of the study drug. Clinically insignificant thrombosis, such as non-obstructive biliary tract-related clots, is not an exclusion criterion. Any history of myocardial infarction, severe/unstable angina, NYHA class 2 or higher heart failure, or left ventricular ejection fraction (LVEF) < 50% on echocardiography, stroke, transient ischemic attack, coronary or peripheral artery bypass surgery, or any acute coronary syndrome, clinically significant supraventricular or ventricular arrhythmias, and symptomatic congestive heart failure within 6 months prior to the first dose of the study drug. Uncontrolled moderate-to-severe hypertension (SBP > 180 mmHg or DBP > 100 mmHg). Poorly controlled arrhythmias (including QTcF interval ≥ 470 ms for females); abnormal corrected QT interval (QTcF) on electrocardiogram (ECG) at rest during screening, with QTcF ≥ 470 ms for females on average of three ECGs taken at least 5 minutes apart. Pericarditis/clinically significant pericardial effusion.Cardiomyopathy.

* Presence of active autoimmune disease or immunodeficiency, including but not limited to autoimmune hepatitis, interstitial pneumonia, uveitis, rheumatoid arthritis, inflammatory bowel disease, hypophysitis, vasculitis, nephritis, etc.
* Pregnant or lactating women, or women of childbearing potential who are unwilling or unable to use effective contraceptives (applicable to both male and female subjects) until at least 6 months after the last trial treatment, confirmed by blood or urine HCG testing.
* Uncontrolled diabetes (referring to large fluctuations in blood glucose despite standard insulin therapy and frequent blood glucose monitoring, affecting the patient's life and frequent occurrences of hypoglycemia).
* Subjects with unsatisfactory asthma control despite systemic treatment with bronchodilators.
* Subjects who have undergone or plan to undergo solid organ or hematological system transplants during the study period (excluding corneal transplants).
* Currently participating in an interventional clinical study treatment or having received other trial drugs or study devices within 4 weeks prior to the first dose; subjects who have not fully recovered from toxicity and/or complications resulting from any intervention prior to the first dose.
* Abnormal coagulation function (INR > 1.5 or prothrombin time [PT] > ULN + 4 seconds or APTT > 1.5 ULN), bleeding tendency, or ongoing thrombolytic or anticoagulant treatment.
* History of psychoactive drug abuse that cannot be discontinued or presence of psychiatric disorders.
* Subjects with genetic or acquired bleeding disorders or coagulation dysfunction (eligibility based on investigator's judgment).
* History of cerebrovascular accident or transient ischemic attack within 6 months.
* Conditions that increase the risk associated with participating in the study or the study drug and, in the investigator's judgment, render the patient unsuitable for enrollment.
* Other conditions deemed unsuitable for participation in the study by the investigator.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 140 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2029-04-01 (Estimated); Study Completion 2029-04-01 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | 36 months
  The time from randomization until tumor progression (as defined by RECIST 1.1 criteria) or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Overall survival, OS | 36 months
  The time from randomization until death from any cause. For subjects who are lost to follow-up before death, the last follow-up time is usually counted as the time of death.
Objective response rate, ORR | 36 months
  The proportion of patients whose tumor volume decreases by a predetermined amount and maintains this reduction for the minimum required duration. It is the sum of the complete response (CR) and partial response (PR) rates. In other words, ORR = CR + PR.
Disease control rate, DCR | 36 months
  The percentage of evaluable patients who achieve a response (PR + CR) or stable disease (SD) after treatment. Simply put, DCR = CR + PR + SD, according to the RECIST criteria for at least 4 weeks.
Duration of Overall Response, DOR | 36 months
  The time from when a patient first achieves a CR or PR to disease progression.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital (PUMCH), Chinese Academy of Medical Sciences, Beijing, China, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Sharing research findings through article publication
Supporting Information: Study Protocol, CSR